CLINICAL TRIAL: NCT06345040
Title: The Dialogue Study: A Randomized Clinical Trial Investigating the Effect of a Virtual-reality Based Treatment for Eating Disorders
Brief Title: The Dialogue Study: A Virtual-reality Based Treatment for Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-22067692
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa
Keywords: Virtual reality-assisted therapy; Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; eating disorder voice; anorexic voice; avatar therapy; externalization; relational therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual-reality assisted therapy + treatment as usual (Experimental): Seven sessions
  Interventions: Behavioral: Virtual-reality intervention
- Treatment as usual (TAU) (Active Comparator): Seven sessions
  Interventions: Behavioral: TAU - specialized treatment

INTERVENTIONS:
Behavioral: Virtual-reality intervention — For the experimental condition, participants will receive seven individual sessions of Virtual Reality Therapy conducted by a therapist trained in both eating disorder psychotherapy and virtual reality-based therapy, including avatar therapy. In the initial stage of therapy participants create a virtual avatar embodying their eating disorder voice. This enables the person to engage in real time face to face dialogue with the eating disorder voice. The main goal of the intervention is to encourage participants to stand up to the negative comments and commands made by the eating disorder voice and hereby increase their power and agency in the context of the eating disorder voice.
  Arms: Virtual-reality assisted therapy + treatment as usual
Behavioral: TAU - specialized treatment — The control condition encompasses treatment as usual comprising seven sessions of specialized treatment, such as individual or group psychotherapy and dietary guidance, provided by interdisciplinary health professionals.
  Arms: Treatment as usual (TAU)

SUMMARY:
The Dialogue Study is a randomized, assessor-blinded parallel-groups superiority clinical trial fulfilling the CONSORT criteria for non-pharmacological treatment. The aim of the trial is to investigate the effect of a new virtual reality based psychotherapy for eating disorders. A total of 96 participants with a diagnosis of anorexia nervosa or bulimia nervosa will be allocated to either Virtual-reality therapy plus treatment as usual or treatment as usual. All participants will be assessed at baseline and 12- and 24 months post baseline. A stratified block-randomisation with concealed randomisation sequence will be conducted. Independent assessors blinded to the treatment will evaluate outcome. Analysis of outcome will be carried out with the intention to treat principles.

DETAILED DESCRIPTION:
Eating disorders can be defined as pathological eating habits and a tendency to overestimate weight and body shape. It affects at least 7 % of the global population and has profound physical and psychological costs for the affected individual comprising a high risk of relapse and death. Additionally, eating disorders are associated with a significant economic burden in terms of health care costs and lower employment rates.

There is considerable interest in the development of novel psychological interventions for eating disorders which are more effective and which target characteristics that could potentially serve as maintaining factors in eating disorder pathology. The majority (94%) of patients with an eating disorder report experiencing a dominant critical internal voice commenting on weight and self-worth, often referred to as the eating disorder voice.

Within psychotic disorders, a virtual reality-based therapy termed avatar therapy has proven highly effective in reducing the power of the psychotic voice and consequently alleviating the associated distress. Building on this evidence we have developed a modified version of the avatar treatment protocol targeting patients with an eating disorder.

The objective of the Dialogue Study is to identify whether this virtual reality-based therapy can reduce symptoms, improve quality of life, and be cost-effective in treating patients with an eating disorder. Two feasibility studies have found the intervention to be feasible and acceptable for individuals with an eating disorder. Evidence on the efficacy of the intervention now needs to be tested in a large methodological rigorous trial. If the results of the randomized clinical trial are positive, it may motivate scalability and potential implementation in the clinics treating adults with an eating disorder.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ Age 18 of years
2. Ability to give informed consent
3. A diagnosis of eating disorder (ICD-10 code: F50.0 - F.50.3)
4. Recognizing having an internal eating disorder voice

Exclusion Criteria:

1. Unable to identify an internal eating disorder voice
2. Organic brain disease
3. Comorbid psychosis
4. Psychotic depression
5. Active suicidal ideations
6. Risk of refeeding syndrome
7. A command of spoken Danish or English inadequate for engaging in therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Eating disorder symptoms post treatment measured with the Eating Disorder Examination Questionnaire | Baseline, at 12 weeks, and at 24 weeks follow up.
  The primary outcome of the study is eating disorder symptoms measured with the Eating Disorder Examination Questionnaire (EDE-Q) post treatment (12 weeks follow up). The EDE-Q is a widely used and validated self-report questionnaire to assess eating disorder psychopathology and behaviors . It comprises 22 items, rated according to a seven-point forced-choice format (0-6). The questionnaire provides information about eating disorders' central behavioral features (e.g., binge eating, vomiting, laxative misuse), with higher scores reflecting greater symptom severity or frequency. There are four subscales: restraint, eating, shape, and weight concern. Cronbach's α = 0.860.

SECONDARY OUTCOMES:
Level of depressive symptoms post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of depressive symptoms post treatment measured with The Hospital Anxiety and Depression Scale (HADS), subscale Depression. HADS is a self-reporting questionnaire consisting of 14 items measuring the level of anxiety and depression. Items for anxiety and depression are scored separately on a scale from 0-3 with a score range of 0-21 for both subscales. The higher the score the higher symptom load.
Motivation for change post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Motivation for change as experienced by the participant post treatment measured with the Stages of Change in Eating Disorders Questionnaire (SOCQ-ED) The SOCQ-ED comprises 13 items measuring motivation to change. For each item, the participant selects among seven different response options which reflects the possible stage of change (i.e. precontemplation, contemplation, preparation, action, maintenance, and termination). Items are rated on a 6-point Likert scale ranging from 1-7, one being the possibility to exclude an irrelevant symptom domain. The higher score the more motivation to change.
Level of identification with the eating disorder and level of embodiment post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of identification with the eating disorder and level of embodiment post treatment measured with the Identity and Eating Disorder Questionnaire (IDEA). IDEA is a 23 item self-report questionnaire assessing identification with the eating order and the experience of being (dis)embodied. Items are rated on a 5-point Likert scale ranging from 0 (do not agree) to 4 (strongly agree). The total score is the average of all item ratings. The higher score the more identification with the eating disorder and the less experienced embodiment.
Experience of the eating disorder voice post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  The experience of the eating disorder voice post treatment assessed with the Experience of An Anorexic Voice Questionnaire (EAVE-Q). The EAVE-Q is a self-report questionnaire containing 18 items covering the experience of the eating disorder voice. Each question is scored from 1 (strongly disagree) to 5 (strongly agree). Higher EAVE-Q score is associated with higher symptom load in terms of eating disorder symptoms, depression- and anxiety symptoms, and decreased quality of life.
Beliefs about the power and benevolence of the eating disorder voice post treatment - engagement scale | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of engagement with the eating disorder voice post treatment measured with the Revised Beliefs About Voices questionnaire (BAVQR), subscale Engagement. BAVQR is a self-report questionnaire with 5 subscales assessing the individual's beliefs about the power and the benevolence/malevolence of the voice and the emotional, and behavioral ways of responding to it. Participants indicate responses on a 4-point Likert scale ranging from disagree (0) to strongly agree (3). The Engagement subscale is divided into emotional and behavioral ways of reacting. The higher score the more emotional and behavioral engagement.

OTHER OUTCOMES:
Total score of eating disorder voice characteristics post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Total score of eating disorder voice characteristics post treatment assessed with a modified version of the Psychotic Symptoms Rating Scale, Auditory Hallucinations (the subscale: PSYRATS-AH). PSYRATS-AH consists of interviewer administered scales on frequency and duration of auditory hallucinations as well as scales on degree of distress associated with them. The modified version assesses frequency and duration of the eating disorder voice as well as the associated distress. Each item is rated on 5-point scale (0-4). The total score of PSYRATS-AH ranges from 0-44 with higher scores reflecting higher frequency, duration and distress.
Level of quality of life post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of quality of life measured with the Eating Disorder Quality of Life Scale (EDQLS). EDQLS measures 12 domains of eating disorder related quality of life (i.e., disease-specific quality of life). Consists of 40 items, each rated on a 5-point Likert scale from strongly disagree (1) to strongly agree (5). Higher scores indicating better/higher ED-related quality of life.
Perceived difference in power between eating disorder voice and eating disorder patient post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Perceived difference in power between eating disorder voice and eating disorder patient post treatment measured with the Voice Power Differential Scale (VPDS). VPDS is a self-report questionnaire with seven items measuring the perceived difference in power between the voice and the voice hearer. Power components include power, strength, confidence, respect, ability to cause harm, superiority, and knowledge. Each component is rated on a 5-point scale (1-5). The higher score, the more power the voice is perceived to have compared to the voice hearer.
Level of acceptance of and action in relation to the eating disorder voice post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of acceptance and action in relation to the eating disorder voice measured with the Voices Acceptance Scale (VAAS). VAAS is a self-reporting 31 item questionnaire comprising three scales: Acceptance, Action, and a full scale. Responses are provided on a 5-point Likert scale ranging from strongly disagree (0) to strongly agree (4) with higher scores meaning higher levels of acceptance and action in relation to the eating disorder voice.
Level of self-compassion post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of self-compassion post treatment measured with The Self-Compassion Scale (SCS). SCS is a 26 item self-report measure examining how individuals typically treat themselves when they are struggling. It consists of 6 subscales (Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, Over-Identification). Participants indicate, on a 5-point Likert scale ranging from Almost Never (1) to Almost Always (5), how often they think and feel as described. Higher scores indicate greater self-compassion.
Level of body dissatisfaction post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of body dissatisfaction measured with the Body Shape Questionnaire (BSQ-34) post treatment: BSQ-34 is a 34 item self-report questionnaire measuring body dissatisfaction, including concerns about body shape. Body dissatisfaction is assessed across four dimensions: avoidance and social shame related to body exposure, dissatisfaction with the lower parts of the body, use of laxatives and vomiting to reduce body dissatisfaction, and cognitions and maladaptive behaviors to control weight. Questions are answered on a Likert scale ranging from never (1) to always (6). Higher scores indicate greater concern about body shape and greater body dissatisfaction.
Level of perceived self-efficacy post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of perceived self-efficacy post treatment measured with the General Self-Efficacy Scale (GSE). GSE consists of 10 items rated on a Likert scale ranging from 1 (not at all true) to 4 (exactly true). Higher scores indicate greater self-efficacy.
Ability to regulate emotion post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Ability to regulate emotion post treatment measured with the Emotion Regulation Questionnaire (ERQ). ERQ is a 10 item self-report questionnaire measuring how the respondent controls (regulates and manages) their emotions in two different ways: Emotional experience (cognitive reappraisal) and emotional expression (expression suppression). Items are answered on a 7-point Likert scale ranging from 1 (completely disagree) to 7 (completely agree). The two subscales are scored separately. Higher scores indicate greater use of the specific emotion regulation strategy.
Level of executive functioning post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of executive functioning post treatment measured with Behavior Rating Inventory of Executive Functioning (BRIEF). BRIEF is a 75 item self-report measure assessing executive functions. Participants indicate whether a specific behavior is a problem on a 3-point Likert scale (0 = Never, 1 = Sometimes, 2 = Often). The global score (General Executive Function) ranges from 0-225. Higher scores indicate more problems with executive functioning.
Participant satisfaction | 12 weeks follow up.
  Participant satisfaction measured with the Client Satisfaction Questionnaire (CSQ). CSQ is an 8 item self-report measure on satisfaction. Responses are given on a 4-point Likert scale ranging from bad (1) to excellent (4). Higher scores indicate higher satisfaction.
Presence of childhood traumas | Baseline.
  Presence of childhood traumas measured with the Childhood Trauma Questionnaire (CTQ). CTQ is a 28 item self-reporting instrument for retrospective assessment of trauma. Answers are given on a 5-point Likert scale ranging from never (1) to very often (5). Higher scores indicates greater severity of childhood trauma.
Level of simulator sickness | 2 weeks and 7 weeks post baseline.
  Level of simulator sickness measured with the Simulator Sickness Questionnaire (SSQ). SSQ is a 16 item self-report measure for simulator sickness. Participants are asked to rate symptoms on a 4-point Likert scale (0-3). The higher score the more symptoms (administered in therapy).
Level of dysfunctional cognitive beliefs post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of dysfunctional cognitive beliefs measured with the Dysfunctional Attitude Scale questionnaire (DAS-24). DAS-24 is a 24 item self-report measure on dysfunctional cognitive beliefs. Responds are given on a 7-point Likert scale ranging from totally disagree (1) to totally agree (7). Higher scores reflect higher levels of dysfunctional beliefs.
Positive and negative aspects of eating disorders as perceived by the participant post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Positive and negative aspects of eating disorders post treatment as perceived by the participant measured with the Pros and Cons of Eating Disorders questionnaire (P-CED). P-CED is a 62 item self-report questionnaire assessing the participants perception of the pros and cons of the eating disorder. Answers are given on a 5-point Likert scale ranging from strongly agree (1) to strongly disagree (5). The sum of the pros and cons respectively are used to form an Ambivalence Score indicating the weight between the two.
Personal recovery post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of personal recovery post treatment measured with the Questionnaire about Process of Recovery (QPR-15)(53). QPR-15 is a 15 item self-report measure for determining the level of personal recovery. Answers are given on a 5-point Likert scale ranging from strongly disagree (0) to strongly agree (4). The higher score the higher level of perceived recovery.
Presence of comorbidity | Baseline.
  Presence of comorbidity at baseline assessed with the Mini International Neuropsychiatric Interview (MINI). MINI is a structured diagnostic interview for the main psychiatric Axis-I diagnoses in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) and International Classification of Diseases, Tenth Revision (ICD-10). Participants are asked questions on mental health problems that require a YES or NO answer. Interviewer based rating is done by marking either YES or NO for each symptom within in each diagnosis module. At the end of each module, there are diagnostic boxes indicating whether the diagnostic criteria are met or not.
Cost effectiveness of the intervention | Baseline, at 12 weeks, and at 24 weeks follow up.
  Analysis of the cost effectiveness of the intervention using the EuroQol Research Foundation self-report questionnaire on health (EQ-5D). EQ-5D asks participants to classify their own health according to five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated according to three levels: no problems, moderate problems or extreme problems defining 243 potential health states.
Level of cognitive (in)flexibility post treatment | Baseline, at 12 weeks, and at 24 weeks follow up.
  Level of cognitive (in)flexibility measured with the Detail and Flexibility Questionnaire in Eating Disorders (Dflex). Dflex is a 24 item self-report questionnaire developed to measure two cognitive thinking styles often reported in patients with an eating disorder: cognitive rigidity (inflexibility) and excessive attention to details. It contains two subscales: Cognitive Rigidity Subscale and Attention to Detail Subscale. Participants respond on a 6-point Likert scale ranging from Strongly Disagree (1) to Strongly Agree (6). The higher the score, the more rigidity/attention to detail.
Monitoring and reporting of adverse and unwanted events | 12 weeks follow up.
  Monitoring and reporting of adverse and unwanted events from psychotherapy measured with the Negative Effects Questionnaire (NEQ). NEQ is a 32 item self-report questionnaire examining events and outcomes that negatively impact the participant (these can be related to circumstances in the individual's life as well as related to treatment). For each item, the participants indicate whether they experience the statement (yes/no). If yes, the participant rates how negatively the event/outcome affected them on a 5-point Likert scale from 0 (not at all) to 4 (very much). Then it is indicated whether the negative event/outcome is related to treatment or other circumstances. The higher score the more negative effects.
Level of immersion in virtual reality | 2 weeks and 7 weeks post baseline.
  Level of immersion in virtual reality (VR) measured with a modified version of the Multi Modal Presence Scale (MPS). MPS modified version is a 10 item self-report scale measuring the level of immersion in VR, relevant to the dialogue intervention's virtual environment. Answers are given on a 5-point Likert scale ranging from totally disagree (1) to totally agree (5). The higher score the more immersion.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Research Center for Mental Health - CORE, Hellerup, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen NK, Ries ES, Ward T, Cardi V, Christensen AB, Hjorthoj C, Nordentoft M, Micali N, Glenthoj LB. The Dialogue study: Protocol for a randomized clinical trial evaluating the efficacy of virtual reality-based psychotherapy plus treatment as usual versus treatment as usual for eating disorders. PLoS One. 2025 Jul 28;20(7):e0319875. doi: 10.1371/journal.pone.0319875. eCollection 2025. PMID 40720536